CLINICAL TRIAL: NCT05131867
Title: Management of Cerebral Vascular Spasm in Posttraumatic Subarachnoid Hemorrhage Using Combination Therapy of Oral Nimodipine and Intravenous Milrinone: Randomized Clinical Trial
Brief Title: Management of Cerebral Vascular Spasm in Posttraumatic Subarachnoid Hemorrhage Using Combination Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, lecture of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6919
Record Dates: First submitted 2021-07-07; First posted 2021-11-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Oral Nimodipine; Milrinone; Vascular Spasm After Traumatic Subarachnoidhaemorrhage
Keywords: milrinone Oral Nimodipine
MeSH Terms: interventions — Nimodipine; Milrinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- triple H group (Active Comparator): The patients will receive nimodipine (60 mg/4 hours) orally or via nasogastric tube from the first day of admission, then after the diagnosis of vasospasm is confirmed, Triple H therapy (hypertension, hypervolemia and hemodilution) will be started. norepnnephrine (0.01-0.2ug/kg/min) to mentain main arterial blood pressure >100mmhg and hypervolemia to maintain the CVP around 12---14 mmHg and hemodilution to maintain the haematocrit between 30% and 33%.
  Interventions: Drug: nimodipine
- Milrinone group (Active Comparator): The patients will receive oral Nimodipine (60 mg/4) will be given orally or in the gastric tube also from the first day of admission, then after the diagnosis of vasospasm is confirmed, start milrinone bolus of 0.1-0.2 mg/kg followed by 0.75mcg/k/min, if no response after 30min increase the infusion to 1-25mcg/kg/min with maintaining CVP 5:8.
  Norepinephrine (0.01-0.2ug/kg/min) is used only to restore the mean arterial pressure (MAP) to its previous values If there was no recurrence of symptoms after 72 h, we decreased the milrinone infusion by 0.25 mcg/kg/min every 24 or 48 h until discontinuation. If there are any recurrent of symptoms of vasospasm, the patients are placed back on the dose they were previously receiving. If required, another Milrinone bolus is administered if the patient's deficits do not revert12.
  Interventions: Drug: Oral Nimodipine and milrinone

INTERVENTIONS:
Drug: nimodipine — (60 mg/4 hours) orally or via nasogastric tube
  Arms: triple H group
Drug: Oral Nimodipine and milrinone — Oral Nimodipine then after the diagnosis of vasospasm is confirmed, start milrinone bolus
  Arms: Milrinone group

SUMMARY:
To evaluate the efficacy and safety of oral Nimodipine and IV milrinone combination therapy for management of cerebral spasm after aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double-blind manner into 2groups each one containing 15 patients.

Group 1(n =15 ):the patients will receive nimodipine (60 mg/4 hours) orally or via nasogastric tube In group 2(n =15 ): the patients will receive Oral Nimodipine (60 mg/4) will be given orally or in the gastric tube also from the first day of admission, then after the diagnosis of vasospasm is confirmed, start milrinone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to our surgical ICU
* aged between (18-60) years old
* World Federation of Neurological Surgeons grades 1-3 Grades

Exclusion Criteria:

* Aneurysmal SAH
* SAH with Fisher Grade I and IV,
* World Federation of Neurological Surgeons grade IV & V
* No informed consent,
* peripheral vascular disease
* Cardiac disease (heart block, severe valvular stenosis, cardiomyopathothy , ejection fraction<40%), Renal impairment (serum creatinine ≥ 1.4 mg.L-1), Hemodynamic instability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Concentration of transcutaneous cerebral mixed oxygen saturation | every 24 hours up to 1 week
  by forehead bilateral interconnected adhesive probes

SECONDARY OUTCOMES:
Number of participants having cerebral infarction (cerebral infarction incidence) | every 48 hours up to 1 week
  detected by computed tomography
Number of participants restore of the previous conscious level and motor state(Percentage of drug success) | 1 hour after administration of milrinone and 2 hours after administration of triple H therapy
  restore of the previous conscious level and motor state
value of Glasgow coma scale | every 24 hours up to total days of ICU and hospital stay
  with minimum scale vlue of 3 is the worst and maximum value of 16 indicate better outcome
Number of participants develop one of adverse events | after administration of the study drugs up to 30 days
  hypotension ,bradycardia,hypotesion
Total ICU and hospital stay | up to 30 days after administration of the study drugs
mortality rate | 30 day after administration of the study drugs
  Number of participants died within 30 day after administration of the study drugs
value of Modified Rankin scale | 3,6,12 monthes after drug administration
  Level 0: no symptoms Level 1: no significant disability, despite symptoms; able to perform all usual duties and activities Level 2: slight disability unable to perform all previous activities but able to look after own affairs without assistance Level 3: moderate disability; requires some help, but able to walk without assistance.
  Level 4: moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance Level 5: sever disability; bedridden, incontinent and requires nursing care and attention
Glasgow Outcome Scale | 3,6,12 monthes after drug administration
  1. Dead: As a direct result of brain trauma, or … due to secondary complications or other complications" "2. Vegetative State: Patients who remain unresponsive and speechless…." "3. Severe Disability: The The patient is conscious but needs the assistance of another person for some activities of daily living every day.…." "4. Moderate Disability: Such a patient is able to look after himself at home, to get out and about to the shops and to travel by public transport. However, some previous activities, either at work or in social life, are now no longer possible by reason of either physical or mental deficit…." "5. Good Recovery: This indicates the capacity to resume normal occupational and social activities, although there may be minor physical or mental deficits…social outcome should be included in the assessment here, such as leisure activities and family relationships..

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Aculty of Medicine,Zagazig University, Zagazig, Sharqia Province
  - Faculty of Medicine,Zagazig University, Zagazig, Zagazig, Elsharkia,egypt

IPD SHARING:
Plan to Share IPD: No